CLINICAL TRIAL: NCT05474287
Title: Hypoxemia During Deep Sedation for Gastrointestinal Endoscopy at High Altitudes: High-flow Nasal Oxygen Therapy vs. Supraglottic Jet Oxygenation and Ventilation
Brief Title: SJOV vs. HFNO for Hypoxia During Procedural Sedation at High Altitudes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chair of Department of Anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XZ2022ZR-ZY11-Z
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Hypoxia; High Altitude
MeSH Terms: conditions — Hypoxia; Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraglottic jet oxygenation and ventilation (Experimental): Supraglottic jet oxygenation and ventilation is conducted for the participants during sedation.
  Interventions: Procedure: SJOV
- High-flow nasal oxygen therapy (Active Comparator): High-flow nasal oxygen therapy is conducted for the participants during sedation.
  Interventions: Procedure: HFNO

INTERVENTIONS:
Procedure: SJOV — SJOV is conducted using a Wei nasal jet tube (WNJ, Well Lead Medical Co. Ltd, Guangzhou, China) which is connected to a manual jet ventilator (Well Lead Medical Co. Ltd, Guangzhou, China) via its jet port. The initial settings of SJOV were as follows: driving pressure (DP) 15 psi; respiratory rate (RR) 20 bpm; inspiratory-to-expiratory (I/E) ratio 1:2, and gas supply, 100% oxygen.
  Arms: Supraglottic jet oxygenation and ventilation
Procedure: HFNO — HFNO is conducted. Oxygen supplementation is delivered at 35 liters min-1 with a fraction of inspired oxygen (FiO2) of 100%.
  Arms: High-flow nasal oxygen therapy

SUMMARY:
This study aims to compare the effect of the use of supraglottic jet oxygenation and ventilation (SJOV) with high-flow nasal oxygen therapy (HFNO) on reducing the rate of hypoxia during gastrointestinal endoscopic procedures in deeply sedated patients at high altitudes.

DETAILED DESCRIPTION:
The participants will be randomly allocated to either SJOV or HFNO in a 1:1 ratio using block randomization with variable block sizes of four or six randomized. In the HFNO group, oxygen supplementation is delivered at 35 liters min-1 with a fraction of inspired oxygen (FiO2) of 100%. In the SJOV group, SJOV is conducted using a Wei nasal jet tube (WNJ, Well Lead Medical Co. Ltd, Guangzhou, China) which is connected to a manual jet ventilator (Well Lead Medical Co. Ltd, Guangzhou, China) via its jet port. The initial settings of SJOV were as follows: driving pressure (DP) 15 psi; respiratory rate (RR) 20 bpm; inspiratory-to-expiratory (I/E) ratio 1:2, and gas supply, 100% oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. underwent routine gastrointestinal endoscopy under procedural sedation;
3. consented to participate in this trial.

Exclusion Criteria:

1. infection of the upper airway;
2. anatomical abnormalities of the face, nose, and upper airway;
3. coagulopathies;
4. anticipated or known difficult airway;
5. known allergy against propofol, soybeans, and egg;
6. absence from the high-altitude environment during the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Hypoxia during sedation | During sedation procedure
  An SPO2 of 75 - 89% for < 60 s

SECONDARY OUTCOMES:
respiratory-related complications | During sedation procedure
  pulmonary aspiration, respiratory depression (SPO2 = 90-95%) and severe hypoxia (SPO2 < 75% or < 90% for > 60s)
cardiovascular-related complications | During sedation procedure
  hypotension (systolic blood pressure < 90 mmHg), hypertension (systolic blood pressure > 160 mmHg), bradycardia (heart rate < 50 beats/min), tachycardia (heart rate > 120 beats/min)
fatal complications | from sedation initiation to 20 min after patients are awake
  severe anaphylactic reactions, myocardial infarction, cardiac arrest and death

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, Principal Investigator — Peking University People's Hospital
Locations (1):
- Tibet autonomous region people's hospital, Lhasa, Tibet, China

IPD SHARING:
Plan to Share IPD: No